CLINICAL TRIAL: NCT00149110
Title: "The CHRONOS Study: Can the Sleep-deprivation Induced Antidepressive Effect in Patients With Major Depression be Sustained by Correction of Diurnal Rhythms, Long Term Light Treatment and Duloxetine Treatment?"
Brief Title: Chronos: the Use of Chronobiological Treatment in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillerod Hospital, Denmark (Other)
Collaborators: Eli Lilly and Company (Industry); The County of Frederiksborg (Unknown)
Responsible Party: Klaus Martiny, Psychiatric Research Unit, Hillerod Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-001855-39 Eudra CT number
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Major Depression
Keywords: Sleep deprivation; Exercise; Light therapy; Major depression; Bipolar depression; Sleep-wake cycle
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Deprivation; Motor Activity; Bipolar Disorder | interventions — Phototherapy; Circadian Rhythm; Exercise; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Sleep deprivation in combination with light and duloxetine
  Interventions: Procedure: Sleep deprivation; Procedure: Light therapy; Procedure: Diurnal rhythms; Drug: duloxetine
- B (Active Comparator): Exercise and duloxetine
  Interventions: Behavioral: Exercise; Drug: duloxetine

INTERVENTIONS:
Procedure: Sleep deprivation — 3 days with a normal night between
  Arms: A
Procedure: Light therapy — Daily light therapy for 29 weeks
  Arms: A
Procedure: Diurnal rhythms — Keeping the day-night cycle constant by use of educational measures
  Arms: A
Behavioral: Exercise — Moderate intensity daily exercise for 30 minutes at least
  Arms: B
Drug: duloxetine — 60 mg daily
  Arms: A
Drug: duloxetine — 60 mg daily
  Arms: B

SUMMARY:
The primary objective of the present study is to examine whether the combination of the antidepressant duloxetine and chronotherapeutic methods (including sleep deprivation, light therapy, and maintaining a regular sleep-wake rhythm) in patient with major depression, will induce an immediate improvement from depression and whether this antidepressive effect will be maintained in the long term (29 weeks). Patient will be randomised to the above mentioned treatment or to an active group receiving exercise.

DETAILED DESCRIPTION:
Protocol synopsis

Background:

The Psychiatric Research Unit at Frederiksborg General Hospital, with professor Per Bech as the driving force, has been working with sleep in relation to affective disorders for many years. During the last 4 years we have performed and been involved in several light therapy studies in depression, both in seasonal affective disorder (SAD), with light as an augmentation strategy in nonseasonal depression, in post-stroke depression and in Tourette's syndrome.

In relation to the dissemination of results from Klaus Martiny's Ph.D. thesis on bright light therapy as an augmenting strategy in major depression, our research unit has achieved close collaboration with some of the world's leading experts in chronotherapeutics: Professor Anna Wirz-Justice in Basel, Switzerland, Franscesco Benedetti in Milano, Italy, Michael Terman in New York, Mathias Berger in Freiburg, Germany and Joseph Wu at the University of California, Irvine. The basic idea of the present study comes from this group which over many years has performed and reported clinical studies in chronotherapeutics. We hope that our research unit will be able to conduct this study, as required, in a large patient sample and under the guidance of this group.

The study will fulfill the research unit's ambition to investigate antidepressive treatment algorithms with the propensity to lead to an earlier and sustained onset of action and a higher remission rate. Remission from depression does not only restore the patients' normal social functioning, but also reduces the risk of recurrence of depression. To attain this goal we regard the combination of new and powerful antidepressive drugs and non-pharmacological therapies most interesting and promising. This study has full support from the hospital administration who welcomes the active involvement of the nursing staff in the chronotherapeutic part.

The present study incorporates the combination of duloxetine and chronotherapeutics: sleep deprivation, sleep phase advance, and light therapy.

Duloxetine is a new dual action antidepressant drug that has shown an early onset of action and a high remission rate, with acceptable side effects. It is thus a promising drug for new studies.

Chronotherapeutic approaches such as total or partial sleep deprivation, phase advance of the sleep-wake cycle, and light therapy have been investigated over the last thirty years.

Total or partial sleep deprivation in the second half of the night and phase advance of the sleep-wake cycle have shown to have rapid and profound effects on depressed mood in all diagnostic subgroups. Sleep deprivation attains an immediate response in around 60% of the cases and smaller reported studies using combinations of sleep deprivation with lithium, antidepressant drugs, pindolol, sleep phase advance, or morning light therapy have indicated that the response after initial sleep deprivation can be maintained. Light treatment has become an accepted and effective treatment of seasonal affective disorder (SAD), and recent studies have document accelerated and augmented response in non-seasonal, and even in chronic depression,as adjunctive treatment to medication.

The combination of the effect of chronotherapeutics and new powerful antidepressant drugs thus is a very interesting and promising approach. While light treatment is widely used, sleep deprivation and sleep phase advance are therapies that are in need of studies with sufficient numbers of patients to evaluate their applicability and efficacy.

Objectives:

Duloxetine, a new dual action drug, has shown promising efficacy with an early onset of action and a high remission rate both in short- and long-term treatment. Thus, Raskin found an impressive remission rate of 50.8% after six weeks and 81.8% after 52 weeks of treatment. The primary objective of the present study is to examine whether the combination of duloxetine and chronotherapeutic methods induces higher remission rates at an earlier time point and obtains a 50% percent remission rate after three weeks of treatment.

Study design:

The study will be a randomised controlled, semi-blind (rater-blind) trial with a fixed dosage trial length of nine weeks. Within this nine weeks period study drugs will be given at a dose of 60 mg duloxetine. Patients will be randomized and start medication with duloxetine one week before starting the chronotherapeutic intervention. This is a precaution not to cause any distress in patients (as could be expected with new possible side-effects and the chronotherapeutic intervention introduced at the same time). The following chronotherapeutic intervention covers one week (seven days) where patients will be admitted to an open ward. If improved sufficiently patients can be discharged at this time point.

Subsequently patients will be seen monthly in an uncontrolled follow-up period ending with a last visit at 6 month after inclusion into the study. In this follow-up period starting from week nine, patients will have the opportunity to alter dosage of study drug or to shift into other medication. The only intervention in this follow up period will be to encourage the patients to keep the daily time structure as instructed during their admittance to the ward.

Patients randomised to group A will be treated with a combination of duloxetine 60 mg per day for 29 weeks and a chronotherapeutic intervention of one weeks duration (see below). Patients randomised to group B will be treated with duloxetine in a dose of 60 mg per day for 29 weeks and individual exercise instructed by a physiotherapist. Patients will be informed that the two intervention groups are based on different time-structuring regimes. The placebo condition has been chosen to secure an similar expectancy rate in the two treatment conditions.

Group A. Duloxetine treatment with 60 mg per day for 29 weeks plus chronotherapeutic intervention of 1 week duration.

* Duloxetine dosage will be 60 mg daily with the possibility of increasing dosage to 90 or 120 mg at week nine for patients with incomplete response.
* Chronotherapeutic intervention

  1. Light treatment: Light treatment will be given with 10.000 lux for 1 hour, individually timed according to the MEQ score.
  2. Sleep deprivation and sleep phase advance: Sleep will be scheduled as shown below.

     * Day one to two: Total sleep deprivation I
     * Day two to three: from 9 pm to 7 am. Sleep-phase-advance I
     * Day three to four: Total sleep deprivation II
     * Day four to five: from 9 pm to 7 am. Sleep phase advance II
     * Day five to six: Total sleep deprivation III
     * Day six to seven: from 9 pm to 7 am. Sleep phase advance III

Group B. Duloxetine treatment with 60 mg per day for nine weeks plus chronotherapeutic intervention with moderate time structure and exercise of 1 weeks duration.

* Duloxetine dosage will be 60 mg daily with the possibility of increasing dosage to 90 or 120 mg at week nine for patients with incomplete response.

From day seven and on, sleep is regulated according to two rules:

1. Not taking naps in the daytime.
2. Getting out of bed by 8 am at the latest.

Concomitant medication:

Oxazepam is allowed for severe agitation and sleep disturbances (except at days of sleep deprivation) in daily doses as mentioned earlier.

Psychometrics:

The diagnosis of major depression will be made by the Mini International Neuropsychiatric Interview (M.I.N.I.). Severity of depression will be assessed by weekly ratings using the interview-based Hamilton Depression Rating scales (17 and 6 items versions, Bech et al 2000) and the newly developed 6 item self-assessment Hamilton scale. Patients will fill in the Global Rating Scale (Preskorn) daily. Side effects will be monitored weekly by the UKU scale. At baseline, the Morningness Eveningness Questionnaire (MEQ) will be used to calculate the individual timing of light.

Time line:

The study starts in September 2005. The inclusion period is 2 years and data will be published in a 6 months' period thereafter.

Efficacy measures:

Primary outcome criteria will be response and remission. Secondary outcome criteria will be the mean of weekly Hamilton ratings (17-items and 6-items versions).

Tertiary outcome criterion will be the time until discharge.

Regulations:

The study will follow the Good Clinical Practice Guidelines and has obtained approval from the local ethical committee, the Danish Data Protection Agency and the Danish Medicines Agency. Patients will sign informed consent forms after written and oral descriptions of the study.

Safety:

All Events, serious Events, Adverse drug reactions and Suspected Unexpected Serious Adverse Reactions will be reported according to the regulatory authorities' rules. Side effects will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of major depression according to DSM-IV
* Patient with major depression as part of a bipolar disorder should be in adequate mood stabilizing therapy at entry to the study
* Age of 18 or above
* A score on the Hamilton Depression Scale, 17 items version of at least 18

Exclusion Criteria:

* Primary psychotic disorder
* Psychotic depression
* Drug or alcohol abuse
* Severe organic brain disease
* Severe suicidal ideation (a score of 2 or above on the Hamilton Depression Scale, 17-items version)
* Mental retardation
* Pregnancy or lactation period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Hamilton score during the 29 weeks trial | 1 week

SECONDARY OUTCOMES:
Cortisol measurements | 1 week
Depression self rating by the Preskorn scale | 9 month

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Martiny Martiny, MD Ph.D., Principal Investigator — Psychiatric Research Unit, Hilleroed Hospital, Denmark
Locations (1):
- Psychiatric Research Unit, Hilleroed Hospital, Hilleroed, Denmark

REFERENCES:
- [Background] Wirz-Justice A, Benedetti F, Berger M, Lam RW, Martiny K, Terman M, Wu JC. Chronotherapeutics (light and wake therapy) in affective disorders. Psychol Med. 2005 Jul;35(7):939-44. doi: 10.1017/s003329170500437x. PMID 16045060
- [Derived] Martiny K, Refsgaard E, Lund V, Lunde M, Sorensen L, Thougaard B, Lindberg L, Bech P. The day-to-day acute effect of wake therapy in patients with major depression using the HAM-D6 as primary outcome measure: results from a randomised controlled trial. PLoS One. 2013 Jun 28;8(6):e67264. doi: 10.1371/journal.pone.0067264. Print 2013. PMID 23840645
- [Derived] Martiny K, Refsgaard E, Lund V, Lunde M, Sorensen L, Thougaard B, Lindberg L, Bech P. A 9-week randomized trial comparing a chronotherapeutic intervention (wake and light therapy) to exercise in major depressive disorder patients treated with duloxetine. J Clin Psychiatry. 2012 Sep;73(9):1234-42. doi: 10.4088/JCP.11m07625. PMID 23059149